CLINICAL TRIAL: NCT00622531
Title: Utilizing, Studying, Evaluating BNP for Monitoring in Patients With Heart Failure (USE-BNP)
Brief Title: Serial BNP Testing for Heart Failure Management
Acronym: USE-BNP
Status: Terminated | Type: Observational
Why Stopped: Study terminated due to insufficient enrollment
Sponsor: Siemens Healthcare Diagnostics Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CTB-Centaur200603
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Heart Failure
Keywords: heart failure; BNP; natriuretic peptide
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- BNP Open: Subjects treated based on clinical assessment and knowledge of BNP values
  Interventions: Device: BNP assay (Siemens ADVIA Centaur BNP)
- Control: Subjects treated based on clinical assessment alone
  Interventions: Other: hidden BNP value

INTERVENTIONS:
Device: BNP assay (Siemens ADVIA Centaur BNP) — Diagnostic test
  Other Names: Siemens ADVIA Centaur BNP
  Groups: BNP Open
Other: hidden BNP value — no intervention
  Groups: Control

SUMMARY:
The scope of the USE-BNP Trial is to investigate whether knowledge of BNP measurements, in conjunction with clinical assessment, in the outpatient setting can guide the management of therapy in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects must be diagnosed with heart failure and have an abnormal BNP reading.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiology or internal medicine clinics
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2007-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
composite endpoint of all cause mortality, hospitalization due to worsening heart failure and administration of IV drug therapy for worsening heart failure. | 12 months

SECONDARY OUTCOMES:
NYHA classifications in the two treatment groups | 12 months
Quality of life assessments of two treatment groups | 12 months
change in therapy based on BNP usage | 12 months
number of serious adverse events for the two groups | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Denis C Phaneuf, MD, Principal Investigator — Centre Hospitalier de l'Université de Montréal (CHUM) Hôpital Hôtel Dieu; Serge Lepage, MD, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke; Boshara Zakhary, MD, Principal Investigator — Virginia Research Institute; Robert Dupuis, MD, Principal Investigator — Centre de santé et de services sociaux région de Thetford; Lee Marcus, MD, Principal Investigator — The Hudson Valley Heart Center; Thao Huynh, MD, Principal Investigator — McGill University Health Centre (MUHC) Montreal General Hospital; Nadia Giannetti, MD, Principal Investigator — McGill University Health Centre (MUHC) Royal Victoria Hospital; David Markham, MD, Principal Investigator — University of Texas Southwestern Medical Center; Paul Heidenreich, Principal Investigator — Palo Alto VA Health Care System; William Little, MD, Principal Investigator — Wake Forest University Health Sciences; Eric Schaefer, MD, Principal Investigator — NYU Langone Health
Locations (11):
- United States (6):
  - Palo Alto VA Health Care System, Palo Alto, California
  - Bellevue Hospital, New York, New York
  - The Hudson Valley Heart Center, Poughkeepsie, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - Virginia Research Institute, Danville, Virginia
- Canada (5):
  - Centre Hospitalier Universitaire de Sherbrooke, Fleurimont, Quebec
  - Centre Hospitalier de l'Université de Montréal (CHUM) Hôpital Hôtel Dieu, Montreal, Quebec
  - McGill University Health Centre (MUHC) Royal Victoria Hospital, Montreal, Quebec
  - McGill University Health Centre (MUHC) Montreal General Hospital, Montreal, Quebec
  - Centre de santé et de services sociaux région de Thetford, Thetford-Mines, Quebec